CLINICAL TRIAL: NCT06577844
Title: Evaluation of the Contribution of a DEMaterialized VIdeo-pedagogical SUpport in the Care Pathway of Lung Cancer Surgery Patients
Acronym: SUVIDEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCAPHM22_0413
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
Keywords: lung cancer; surgery; anxiety; video support
MeSH Terms: conditions — Lung Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental)
  Interventions: Other: video support
- control (No Intervention)

INTERVENTIONS:
Other: video support — video support provided to the patient before surgery
  Arms: experimental

SUMMARY:
Uni-centric, randomized, open-label, prospective interventional-comparative study, with a control arm (patients receiving standard preoperative information) and an experimental arm (patients receiving standard preoperative information and having access to a dematerialized educational video support).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over,
* Patients requiring surgical management:

for therapeutic purposes (in the case of proven tumor histology) or for diagnostic and therapeutic purposes (in the absence of proven histology, but strong suspicion, after validation by RCP),

- Patients who have given their consent.

Exclusion Criteria:

* Patients under guardianship
* Patients with a history of thoracic surgery
* Patients on long-term analgesic medication
* Patients who do not speak French
* Patients unable to read or write
* Patients with major visual impairment
* Patients with chronic anxiety or depression at the time of admission
* Patients under guardianship
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Immediate pre-operative anxiety | 10 days
  self-measurement using the HAD Scale

SECONDARY OUTCOMES:
Perioperative anxiety (randomization (consultation), immediate postoperative and discharge) | 90 days
  based on HAD scale
Post-traumatic stress disorder | 90 days
  PCL-5 scale
Quality of life evaluation | 90 days
  European Organisation for Research and Treatment of Cancer core health- related quality of life questionnaire (QLQ-C30).
Cumulative postoperative morbidity | 90 days
  score CCI
Intra-hospital consumption of analgesics | 90 days
  accounting for in-hospital consumption of analgesics

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance publique Hopitaux de Marseille - Hopital Nord, Marseille, France

IPD SHARING:
Plan to Share IPD: No